CLINICAL TRIAL: NCT04696159
Title: Impact of Endoscopic Per-Oral Pyloromyotomy (POP) on Glycemic Control in Gastroparesis Patients With Poorly Controlled Diabetes Mellitus
Brief Title: Impact of Per Oral Pyloromyotomy (POP) on Glycemic Control in Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Allemang (Other)
Collaborators: Society of American Gastrointestinal and Endoscopic Surgeons (Other)
Responsible Party: Sponsor-Investigator, Matthew Allemang, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-1460
Record Dates: First submitted 2020-08-14; First posted 2021-01-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus; Gastroparesis With Diabetes Mellitus; Gastroparesis
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis | interventions — Pyloromyotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endoscopic Per-Oral Pyloromyotomy (POP) (Experimental): The study cohort will include 40 patients with a HbA1c >7.5% with medically refractory gastroparesis who are scheduled to undergo POP. Each patient will undergo two 10-day periods of CGM at an interval of approximately seven months, one month prior to the procedure and six months after. Symptoms and diabetes management improvement will be measured by the Gastroparesis Cardinal Symptom Index (GCSI) scores and the Diabetes Self-Management Questionnaire (DSMQ).
  Interventions: Procedure: Pyloromyotomy

INTERVENTIONS:
Procedure: Pyloromyotomy — Endoscopic Per-Oral Pyloromyotomy (POP)

SUMMARY:
This study will assess changes in glycemic control in 40 patients with diabetes who undergo per-oral pyloromyotomy (POP) for medically refractory gastroparesis.

DETAILED DESCRIPTION:
This will be a prospective study using HbA1c values and continuous glucose monitoring (CGM) to assess changes in glycemic control in patients with diabetes who undergo per-oral pyloromyotomy (POP) for medically refractory gastroparesis. The study cohort will consist of 40 patients with poor glycemic control who undergo POP. The investigators propose a prospective cohort study using CGM to compare glycemic profiles before and after POP in patients with diabetic gastroparesis. The investigators hypothesize that patients will have improvement in glycemic control and reduced variation in blood glucose levels (% time in hypo/hyperglycemia) after undergoing POP. These results will aid in clinical decision making, and may indicate an earlier need for endoscopic intervention in patients with uncontrolled diabetes and gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age and older
2. Patients with gastroparesis with an average HbA1c> 7.5% over the past 3 months
3. Patient that have a diagnosis of gastroparesis established by documented delayed gastric emptying by either a wireless motility capsule study or a nuclear gastric emptying study, with no evidence of gastric obstruction.
4. Patients are able to complete all study requirements

Exclusion Criteria:

1. Patients <18 years of age
2. Patients with gastroparesis with an average HbA1c< 7.5% over the past 3 months
3. Patients unable or refuse to complete the study requirements
4. Patients who are unable or refuse to wear a CGM sensor
5. Patients with insulin pumps
6. Patients who already use a CGM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1C levels | Baseline and 6 Month
  Glycemic control will be evaluated by measuring change in Hemoglobin A1C (HbA1c) levels. Poor glycemic control defined as an average HbA1c > 7.5%. Change = (Six Month Score - Baseline Score)
Change from Baseline in Glucose Levels measured by Continuous Glucose Monitor | Baseline and 6 Month
  Glycemic control will be evaluated by measuring average glucose levels using Continuous Glucose Monitors (CGM). Normal glucose levels 74-99 mg/dL. Change = (Six Month Score - Baseline Score)

SECONDARY OUTCOMES:
Change from Baseline on Diabetes Self-Management Questionnaire | Baseline and 6 Month
  The Diabetes Self-Management Questionnaire (DSMQ) is a self reported instrument assessing diabetes self-care activities. Possible scores range from 0 (Does not apply) to 3 (Applies to me very much). Change = (Six Month Score - Baseline Score)
Change from Baseline on Gastroparesis Cardinal Symptom Index | Baseline and 6 Month
  The Gastroparesis Cardinal Symptom Index (GCSI) is a validated patient-administered questionnaire that is used to assess gastroparesis symptom severity. Possible scores range from 0 (None) to 5 (Very Severe). Change = (Six Month Score - Baseline Score)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Allemang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung HK, Choung RS, Locke GR 3rd, Schleck CD, Zinsmeister AR, Szarka LA, Mullan B, Talley NJ. The incidence, prevalence, and outcomes of patients with gastroparesis in Olmsted County, Minnesota, from 1996 to 2006. Gastroenterology. 2009 Apr;136(4):1225-33. doi: 10.1053/j.gastro.2008.12.047. Epub 2008 Dec 24. PMID 19249393
- [Background] Rodriguez J, Strong AT, Haskins IN, Landreneau JP, Allemang MT, El-Hayek K, Villamere J, Tu C, Cline MS, Kroh M, Ponsky JL. Per-oral Pyloromyotomy (POP) for Medically Refractory Gastroparesis: Short Term Results From the First 100 Patients at a High Volume Center. Ann Surg. 2018 Sep;268(3):421-430. doi: 10.1097/SLA.0000000000002927. PMID 30004920
- [Background] Ramzan Z, Duffy F, Gomez J, Fisher RS, Parkman HP. Continuous glucose monitoring in gastroparesis. Dig Dis Sci. 2011 Sep;56(9):2646-55. doi: 10.1007/s10620-011-1810-z. Epub 2011 Jul 7. PMID 21735078
- [Background] Tanenberg RJ, Pfeifer MA. Continuous glucose monitoring system: a new approach to the diagnosis of diabetic gastroparesis. Diabetes Technol Ther. 2000;2 Suppl 1:S73-80. doi: 10.1089/15209150050214168. No abstract available. PMID 11469637
- [Background] Bailey TS, Chang A, Christiansen M. Clinical accuracy of a continuous glucose monitoring system with an advanced algorithm. J Diabetes Sci Technol. 2015 Mar;9(2):209-14. doi: 10.1177/1932296814559746. Epub 2014 Nov 3. PMID 25370149
- [Background] Role of Continuous Glucose Monitoring in Diabetes Treatment. Arlington (VA): American Diabetes Association; 2018 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK538971/ PMID 30958664
- See also: Clinical Guideline: Management of Gastroparesis [Internet]. [cited 2019 Aug 22]. — http://www-ncbi-nlm-nih-gov.ccmain.ohionet.org/pmc/articles/PMC3722580/